CLINICAL TRIAL: NCT02177110
Title: A Translational Systems Medicine Approach to Provide Predictive Capacity for Therapy Responsiveness in Advanced or Metastatic Malignant Melanoma (SYS-ACT)
Brief Title: A Translational Systems Medicine Approach to Provide Predictive Capacity for Therapy Response in Advanced or Metastatic Malignant Melanoma
Acronym: SYS-ACT
Status: Completed | Type: Observational
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: ICORG 13-22
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Advanced Melanoma; Metastatic Melanoma
Keywords: advanced melanoma; metastatic melanoma; fresh frozen tissue; FFPE tissue
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh frozen and FFPE tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study: Patients who have fresh frozen and FFPE tissue taken prior to treatment
- Control: Fresh frozen tissue and FFPE tissue is available

SUMMARY:
This is an exploratory prospective translational multicentre study. Melanoma is the 5th most common cancer diagnosed in Ireland and its incidence among women and men is above the European average.

Following treatment the elimination of cancer cells ultimately occurs by the activation of apoptotic cell death pathways. The SYS-ACT approach builds on a combination of mathematical systems of modelling, quantitative biochemistry and cell biology, and specifically predicts the drug responsiveness of melanoma cell lines to various apoptosis-inducing treatments.

The investigators propose to validate the SYS-ACT approach and application in a translational systems medicine study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age.
2. Patient must be able to give own signed informed consent.
3. Patients that present with advanced or metastatic (stage III/IV) malignant melanoma of the skin.
4. Patients that are planned to receive either:

   * Adjuvant treatment
   * 1st line treatment for metastatic disease
   * 2nd line treatment for metastatic disease
5. Patients with prior adjuvant treatment are allowed.
6. Patients receiving planned standard treatment of one or more of the following:

   * Chemotherapy regimens containing DTIC, TMZ and/or cisplatin
   * Immunotherapy (for example ipilimumab and/or anti-PD-L1/PD-1 therapies)
   * BRAF and/or MEK inhibitors
7. Patients were FFPE and fresh frozen tissue is available (both mandatory).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have a diagnosis of advanced or metastatic melanoma of the skin
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Validation of SYS-ACT | 2 years
  Validate the predictive capacity of SYS-ACT by assessing responsiveness to treatment
Progression free survival | 2 years
  Progression free survival (PFS) and overall survival will be assessed for each patient for up to 2 years.

CONTACTS AND LOCATIONS:
Locations (6):
- Ireland (6):
  - Cork University Hospital, Cork
  - Beaumont Hosptial, Dublin
  - Mater Misericordiae University Hospital and Mater Private Hospital, Dublin
  - St Vincent's University Hospital, Dublin
  - Galway University Hospital, Galway
  - Waterford Regional Hospital, Waterford